CLINICAL TRIAL: NCT06963411
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Crossover Study Evaluating the Safety, Tolerability and Pharmacokinetics of Various Doses of KP001 (Epinephrine Inhalation Aerosol) in Healthy Adult Volunteers While Assessing Carryover Effects
Brief Title: Phase 1 Crossover Study Evaluating the Safety, Tolerability, and Pharmacokinetics of KP001 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kokua Pharma Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP001-101
Record Dates: First submitted 2025-04-24; First posted 2025-05-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Acute Allergic Reaction; Anaphylaxis
Keywords: Epinephrine; Aerosol; Inhalation; Immunotherapy; Upper airway laryngeal edema; Upper airway pharyngeal edema; Hypersensitivity, immediate; Anaphylaxis; Vasoconstrictor agents; Adrenergic alpha-Agonists; Adrenergic beta-Agonists; Bronchodilator agents
MeSH Terms: conditions — Anaphylaxis; Respiratory Aspiration; Hypersensitivity, Immediate

STUDY DESIGN:
Intervention Model Description: The order of the treatment arms A and B will be randomized, all subjects will proceed to Arm C once Arms A and B are completed. Subjects will receive the same treatment they were assigned to in all 3 arms (either KP001 or placebo). There will be a 7-day washout period between the repeated doses of Arms A and/or B, and a subsequent 7-day washout period, once both Arms are completed, when all subjects will be assigned to Arm C. Sequences will be AABBC or BBAAC and carried out as follows:
  AABBC - Treatment A/ 7 day washout/ Repeat Treatment A/ 7 day washout/ Treatment B / 7 day washout/ Repeat Treatment B/ 7 day washout/ Treatment C
  OR
  BBAAC - Treatment B/ 7 day washout/ Repeat Treatment B/ 7 day washout/ Treatment A/ 7 day washout/ Repeat Treatment A/ 7 day washout/ Treatment C.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment Arm A: Two Treatments (Experimental): Subjects will receive two sets of treatments of 0.25 mg (2 inhalations of 0.125 mg each time) of KP001 (or matching placebo) over 2 visits separated by a 1-week washout period. Investigational Product (IP) will be delivered as 1 set of 2 inhalations (2 total) spaced approximately 10 seconds apart.
  Subjects will repeat Arm therefore total dose in mg for Arm = 0.5 mg.
  Interventions: Drug: KP001; Drug: Placebo
- Treatment Arm B: Four Treatments (Experimental): Subjects will receive four sets of treatments of 0.25 mg (2 inhalations of 0.125 mg each time), totaling 1.0mg of KP001 (or matching placebo) over 2 visits separated by a 1-week washout period. IP will be delivered as 4 sets of 2 inhalations (8 total) spaced approximately 10 seconds apart. Each set of 2 inhalations will be spaced approximately 2 minutes apart.
  Subjects will repeat Arm therefore total dose in mg for Arm = 2.0 mg.
  Interventions: Drug: KP001; Drug: Placebo
- Treatment Arm C: Breath Hold (Experimental): Subjects will receive 0.5 mg of KP001 (or matching placebo) delivered as 4 rapidly administered sequential inhalations (4 total), dosed approximately 5 seconds apart, spaced over approximately 15 seconds while holding their breath during the entire dosing treatment and after treatment for a total minimum 30 seconds (or longer) before exhaling.
  Total dose in mg for Arm = 0.5 mg.
  Interventions: Drug: KP001; Drug: Placebo

INTERVENTIONS:
Drug: KP001 — Epinephrine Inhalation Aerosol (0.125 mg per inhalation)
Drug: Placebo — Matched Placebo control (KP001 vehicle only)

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and pharmacokinetics (PK) of several KP001 dose regimens to identify a treatment regimen with a PK profile that safely meets or exceeds the PK profile of existing injected epinephrine products. The main questions it aims to answer are:

* To evaluate any carryover effect with a 7-day washout of different dose regimens of KP001 in healthy adult volunteers.
* To evaluate the safety, tolerability and PK of different dose regimens of KP001 in healthy adult volunteers.
* To explore the safety, tolerability and PK of one KP001 dose regimen without inhalation (breath holding).

Participants will:

* Be admitted to clinical research unit (Day -1) and receive treatment the following day (Day 1) and then will be discharged
* Visit the clinic on Days 2 & 3 post dose for required assessments
* Visit the clinic 6 days post their last dose for dosing and repeated until 5 dosing visits have been completed
* Visit the clinic for a safety follow-up visit approximately 1 week from last dose administered

DETAILED DESCRIPTION:
This study is a 5-period crossover design to evaluate the safety, tolerability, and PK of KP001 compared to placebo and to evaluate for the potential for carryover effect (Arms A & B). An exploratory 3rd arm (Arm C) will evaluate the PK of KP001 when breath holding to replicate an unconscious patient situation, and results will be used to design a possible future breath-holding study. Sequence will be either AABBC or BBAAC. Two doses of KP001 (0.25 mg or 1.0 mg) or placebo will be administered to 16 subjects (12 active and 4 placebo subjects) on two separate occasions, separated by a 1-week washout period. A third arm will evaluate one dose of KP001 (0.5 mg) PK while breath holding.

The total study duration for subjects will be up to 11 weeks, consisting of:

* Participation in up to 6-week screening period
* Attendance of 5 in-patient dosing visits, separated by 1 week
* Attendance of 1-week post-treatment follow up period

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), aged ≥ 18 to ≤ 45 years.
2. A Body Mass Index (BMI) ≥18.5 and ≤ 30 kg/m^2, with body weight, ≥ 50.0 kg for males and ≥ 45.0 kg for females.
3. Healthy as defined by a) the absence of clinically significant illness and surgery within 4 weeks prior to study drug administration. b) the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
4. Normal lung function measured by spirometry.
5. Demonstrated ability to successfully complete pressurized metered dose inhaler (pMDI) training.
6. Demonstrated ability to successfully hold their breath for a minimum of 30 seconds.

Key Exclusion Criteria:

1. Positive urine drug screen, urine cotinine test, or alcohol breath test, at screening.
2. Known reaction or sensitivity to sympathomimetic amines, or idiosyncratic reaction to epinephrine or any of the ingredients of KP001, placebo.
3. History of anaphylaxis or other severe allergic reactions (e.g., angioedema)
4. Surgical procedures within 90 days of admission that could result in confounding of results or additional risk to the subject, per the judgment of the Investigator.
5. History or presence of alcohol abuse or drinking more than 2 standard drinks per day/10 standard drinks per week for women or 3 standard drinks per day/15 standard drinks per week for men; or a positive alcohol breath test at screening or admission.
6. History or presence of drug abuse/dependence (not including nicotine and caffeine) within the previous 1 year or a positive urine drug test at screening or admission.
7. Use of any tobacco or nicotine-containing products within 3 months prior to screening.
8. Use of any inhaled products, including vaping and water pipes (Hookahs) within 6 months prior to screening.
9. Use of any prescription medications within 14 days prior to admission, or over-the-counter medications (including herbal remedies and supplements) within 7 days prior to admission, with the exception of the occasional use of acetaminophen (up to 2 g daily), or an anticipated need to use them during the study.
10. A depot injection or implant of any drug (other than hormonal contraceptives) within 3 months prior to dosing.
11. Monoamine oxidase (MAO) inhibitors within 30 days prior to dosing.
12. Positive test for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBsAg) at screening.
13. Abnormal clinical laboratory findings, vital signs, or ECG
14. Females who are pregnant or lactating, or who have a positive pregnancy test at screening or admission.
15. Donated plasma within 7 days prior to screening, or donation or loss of whole blood (excluding the volume drawn during screening for this study) as follows: 50 to 499 mL of whole blood within 30 days prior to screening, or ≥ 500 mL of whole blood within 56 days prior to screening.
16. Participation in another clinical study involving an investigational drug within 30 days prior to screening, an investigational biologic within 90 days prior to screening, or current/planned participation in another interventional study during this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
The maximal observed plasma concentration (Cmax) | 1 hour pre-dose to 6 hours post-dose on Day 1, 8, 15, 22 and 29
  Blood samples for PK collected at pre dose (-60, -30, -15 mins prior to dosing) and 1, 2, 3, 5, 7, 9, 12, 15, 20, 30, 45, 60, 90 min postdose and, 2-, 6 hours post-dose.
Area under the concentration-time curve from time zero to last measurable concentration (AUC0-t) | 1 hour pre-dose to 6 hours post-dose on Day 1, 8, 15, 22 and 29
  Blood samples for PK collected at pre dose (-60, -30, -15 mins prior to dosing) and 1, 2, 3, 5, 7, 9, 12, 15, 20, 30, 45, 60, 90 min postdose and, 2-, 6 hours post-dose.
Area under the concentration-time curve from time zero to infinity (AUC0-inf) | 1 hour pre-dose to 6 hours post-dose on Day 1, 8, 15, 22 and 29
  Blood samples for PK collected at pre dose (-60, -30, -15 mins prior to dosing) and 1, 2, 3, 5, 7, 9, 12, 15, 20, 30, 45, 60, 90 min postdose and, 2-, 6 hours post-dose.
Time when the maximal plasma concentration is observed (Tmax) | 1 hour pre-dose to 6 hours post-dose on Day 1, 8, 15, 22 and 29
  Blood samples for PK collected at pre dose (-60, -30, -15 mins prior to dosing) and 1, 2, 3, 5, 7, 9, 12, 15, 20, 30, 45, 60, 90 min postdose and, 2-, 6 hours post-dose.
Rate at which drug is removed from the body (Kel) | 1 hour pre-dose to 6 hours post-dose on Day 1, 8, 15, 22 and 29
  Blood samples for PK collected at pre dose (-60, -30, -15 mins prior to dosing) and 1, 2, 3, 5, 7, 9, 12, 15, 20, 30, 45, 60, 90 min postdose and, 2-, 6 hours post-dose.
Half-life of drug (T1/2) | 1 hour pre-dose to 6 hours post-dose on Day 1, 8, 15, 22 and 29
  Blood samples for PK collected at pre dose (-60, -30, -15 mins prior to dosing) and 1, 2, 3, 5, 7, 9, 12, 15, 20, 30, 45, 60, 90 min postdose and, 2-, 6 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Francoeur, MD, Principal Investigator — Syneos HealthClinique Inc.
Locations (1):
- Syneos HealthClinique Inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately after publication, and for a period of 5 years.
Access Criteria: Any purpose. URL to be added.